CLINICAL TRIAL: NCT02033265
Title: Perineural Ultrasound-Guided Axillary Brachial Plexus Block: Influence of Obesity on Block Performance Time, Failure Rate and Incidence of Acute Complications
Brief Title: Ultrasound-Guided Axillary Brachial Plexus Block: Influence of Obesity
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Shalini Dhir, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: IRB00000940
Record Dates: First submitted 2014-01-09; First posted 2014-01-10 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Obesity; Morbid Obesity
Keywords: Ultrasound-guided Axillary Brachial Plexus Block; Obesity; Performance time; Failure rate; Acute complications
MeSH Terms: conditions — Obesity; Obesity, Morbid | interventions — Brachial Plexus Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with BMI less than 30 kg/m2: Patients with BMI less than 30 kg/m2 undergoing surgical procedures on upper limb (elbow, forearm and hand) scheduled to receive ultrasound-guided axillary brachial plexus block as their primary anesthetic modality at SJHC.
  Interventions: Procedure: Brachial plexus block
- Patients with BMI 30 or above: Patients with BMI 30 kg/m2 undergoing surgical procedures on upper limb (elbow, forearm and hand) scheduled to receive ultrasound-guided axillary brachial plexus block as their primary anesthetic modality at SJHC
  Interventions: Procedure: Brachial plexus block

INTERVENTIONS:
Procedure: Brachial plexus block — Ultrasound guided axillary brachial plexus block
  Other Names: Axillary block

SUMMARY:
Axillary brachial plexus block (freezing the nerves in armpit) is commonly performed as a primary anesthetic technique for the elbow/ forearm or hand surgery. These nerves are identified using ultrasound and nerve stimulator (by stimulating the nerves using a small current through the needle). Axillary brachial plexus block has been shown to result in better pain relief, less nausea, vomiting and early discharge from hospital. The use of these nerve blocks have also shown to decrease the duration of hospital stay, decreased side effects of opioids painkillers and better satisfaction scores over the conventional use of intravenous and oral pain medications. These beneficial effects are particularly useful for patients who are overweight or obese. A study by Hauouz et al published in Anesthesia and Analgesia in July 2010 suggests that the success rate of brachial plexus block is lower for obese and overweight patients. However, ultrasound guidance was not used for performing axillary brachial plexus block in this study. We propose that with usage of ultrasound guidance the success rate of brachial plexus block will be similar in obese and non-obese patients.

In this study, we want to compare the success rate of axillary brachial plexus block for obese and non-obese patient groups. We would also like to look at performance time, complications and patient satisfaction for our study population.

DETAILED DESCRIPTION:
The prevalence of obesity is increasing throughout the world. General Anesthesia for obese patients is associated with increased risk of difficult/failed tracheal intubation and aspiration of gastric contents. These life-threatening complications can be avoided by use of regional anesthesia. Other potential advantages of regional anesthesia include improved pain control, less incidence of nausea and vomiting, early ambulation, decreased pulmonary complications, shorter hospital stay. On the other hand, regional anesthesia in obese patients can be challenging because of loss in anatomical landmarks. However, the availability of high-resolution ultrasound imaging has decreased the reliance on anatomical landmarks as the vascular, nervous and musculoskeletal structures can be directly visualized. Ultrasound imaging also allows real time needle visualization and local anesthetic can be deposited more precisely allowing faster onset anesthesia and reduced incidence of complications. Brachial plexus can be anaesthetized at various levels along its course to provide anesthesia for elbow, forearm and hand surgery. Axillary region is ideal site for targeting brachial plexus in obese patients as the plexus is superficial in this region and the likelihood of causing serious complications (e.g. pleural puncture) is low. Study of 188 patients by Chan et al showed that use of ultrasound increases the success rate of axillary brachial plexus block from 63% to 80% when compared with nerve stimulation technique. A recent study (Hanouz et al) showed that obesity increases the failure rate and immediate complications of axillary brachial plexus block but ultrasound was not used for performing the block. In current era, we consider ultrasound-guidance as a standard of care. We hypothesize that the block performance time, success rate and incidence of acute complications are similar in obese and non-obese patients when ultrasound-guidance is used to perform brachial plexus block in axillary region.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgical procedures on upper limb (elbow, forearm and hand) scheduled to receive ultrasound-guided axillary brachial plexus block as their primary anesthetic modality at SJHC
* American Society of -Anaesthesiologists' (ASA) status I to III

Exclusion Criteria:

1. Patients with associated significant cardiac and respiratory disease (ASA status 4/5)
2. Patients with coexisting hematological disorder or with deranged coagulation parameters.
3. Patients with pre-existing major organ dysfunction such as hepatic and renal failure.
4. Psychiatric illnesses
5. Emergency surgery
6. Lack of informed consent.
7. Allergy to any of the drugs used in the study
8. Contraindications to brachial plexus block

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgical procedures on upper limb (elbow, forearm and hand) scheduled to receive ultrasound-guided axillary brachial plexus block as their primary anesthetic modality at SJHC
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Block success rate at 30 minutes | 30 minutes after block performance

SECONDARY OUTCOMES:
Block performance time | Immediate
Incidence of acute complications | Immediate and 48 hours after block performance

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Dhir, FRCPC, Principal Investigator — Lawson Health Research Institute & Western University
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada